CLINICAL TRIAL: NCT04520022
Title: Single Center, Single Group Assignment, Open Label Trial to Assess Safety and Effectiveness of Intravenous Allogeneic Umbilical Cord Blood-derived Mesenchymal Stem Cell in Patients With Recessive Dystrophic Epidermolysis Bullosa
Brief Title: Safety and Effectiveness Study of Allogeneic Umbilical Cord Blood-derived Mesenchymal Stem Cell in Patients With RDEB
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Sang Eun Lee, Assistant professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2015-0285
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: umbilical cord blood-derived mesenchymal stem cell
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FURESTEM-CD Inj (Experimental)
  Interventions: Drug: Human Umbilical Cord Blood-derived Mesenchymal Stem Cells

INTERVENTIONS:
Drug: Human Umbilical Cord Blood-derived Mesenchymal Stem Cells — 3.0 x 106 cells/kg, IV, Total of 3 doses every 2weeks
  Other Names: hUCB-MSCs; FURESTEM-CD Inj

SUMMARY:
Previously, many studies have been conducted on mesenchymal stem cells derived from bone marrow or subcutaneous fat, but interest in cord blood-derived mesenchymal stem cell treatments has been increasing recently.

In the case of cord blood as a source, the isolation of mesenchymal stem cells is easier than bone marrow or fat tissue, and cord blood-derived mesenchymal stem cells have an advantage as a treatment because they have faster population doubling time.

To date, no clinical research on the treatment of patients using cord blood-derived mesenchymal stem cells has been reported in the literature, but there have already been registered at clinicaltrials.gov and currently being conducted overseas.

In this study, we will study the safety and effectiveness of RDEB patient treatment using cord blood-derived mesenchymal stem cells with these advantages.

DETAILED DESCRIPTION:
Until now, all clinical trials for Recessive Dystrophic Epidermolysis Bullosa (RDEB) have examined the potential of bone marrow-derived MSCs. However, umbilical cord blood (UCB) is another important source of stem cells, since its non-invasive collection procedure and rapid availability from cord blood banking. Human UCB-derived MSCs (hUCB-MSCs) exhibit high proliferation capacity and low immunogenicity. A few data support that UCB-MSCs may have significantly greater immunosuppressive potential than other sources of MSCs. A preclinical study has demonstrated that systemic infusions of human UCB-derived unrestricted somatic stem cells, a subpopulation of non-hematopoietic stromal stem cells, significantly extended the life span and reduced blistering of RDEB mice model. Given the promising results of the preclinical study, we conducted a first-in-human, phase 1/2a clinical trial of intravenous administrations of allogeneic hUCB-MSCs in patients with RDEB to determine the safety, tolerability, and potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who diagnosed with recessive dystrophic epidermolysis bullosa through clinical, histological(Partial or complete loss of VII collagen (C7) should be confirmed by DIF and electron microscopy examination) and genetic testing(COL7A1 Genetic mutation must be confirmed).
2. RDEB patients aged 10 to 60 years old (In the case of patients under the age of 19, patients who obtain consent from a representative (parental authority or guardian))
3. Patients who have heard the purpose and contents of a clinical trial and voluntarily signed the consent form prior to the clinical trial (Legal representative in case of minor)
4. Patients who can be monitored during a clinical trial period

Exclusion Criteria:

1. Patients who disagree with this study
2. Patients who is not accompanied by a guardian if those with impaired consent ability
3. Patient or the patient's representative is unable to hear and understand the explanation
4. In case of received immunotherapy or chemotherapy including oral corticosteroid (topical treatment is possible) for more than 1 week within 8 weeks before registration.
5. All kinds of live vaccines except influenza vaccine within four weeks prior to registration
6. Clinically significant infections within four weeks of the screening date or during the screening period (pneumonia, pyelonephritis, Clostridium difficile etc)
7. All kinds of confirmed congenital or acquired immunodeficiency syndrome
8. Acute, chronic infection (Type B, Type C) corresponding to:

   - HBs-Ag, IgM anti-HBc, IgG anti-HBc positive (However, if HBs-Ag and IgM anti-HBc is negative, but only IgG anti-HBc is positive, if ani-HBs Ab positive, this clinical trial can be registered.)
9. Patients who with allogenic stem cell treatment experience within 1 year from the screening test date
10. Patients who have a history of malignant tumors or is currently being treated (squamous cell carcinoma of the skin, cutaneous squamous cell carcinoma inclusion)
11. Type VII collagen ELISA positive and IIF positive
12. Pregnant or lactating women (Women of childbearing potential should agree to use appropriate contraceptive methods (hormonal or barrier method of contraception or abstinence) prior to enrollment in the study and during the study period, including one month after the last administration of the test drug. If pregnant or suspected of being pregnant while participating in the study, the investigator should be informed immediately.)
13. Other cases where the researcher judges that participation in this clinical trial is inappropriate
14. If other clinical trial drugs have been administered within 4 weeks prior to registration or are currently participating in a clinical trial

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Adverse events related to the intravenous allogeneic umbilical cord blood-derived mesenchymal stem cell | 8 months

SECONDARY OUTCOMES:
Change in type VII collagen and anchoring fibril expression at dermoepidermal junction | baseline, day 56
Change in Birmingham Epidermolysis Bullosa Severity Score (BEBSS) | baseline, day56, day 112, day168
Change in Global severity score | baseline, day56, day 112, day168
Change in total body surface area affected by RDEB | baseline, day56, day 112, day168
Change in Quality of Life in Epidermolysis Bullosa (QOLEB) questionnaire | baseline, day56, day 112, day168
Change in blister count | baseline, day56, day 112, day168
Change in pruritus visual analogue scale (VAS) | baseline, day56, day 112, day168
Change in pain visual analogue scale (VAS) | baseline, day56, day 112, day168

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee SE, Lee SJ, Kim SE, Kim K, Cho B, Roh K, Kim SC. Intravenous allogeneic umbilical cord blood-derived mesenchymal stem cell therapy in recessive dystrophic epidermolysis bullosa patients. JCI Insight. 2021 Jan 25;6(2):e143606. doi: 10.1172/jci.insight.143606. PMID 33491668